CLINICAL TRIAL: NCT05837390
Title: Can Cervical Stiffness in the Second Trimester Predict Preterm Birth in High-Risk Singleton Pregnancies?
Acronym: PRECISION
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001714
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Cervical stiffness; cervical integrity
MeSH Terms: conditions — Premature Birth | interventions — FFN protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal swabs.
  Two high vaginal swabs will be obtained as gifted samples for future research. These vaginal swab samples will be stored as part of the LWH tissue bank for 2 years for future exploratory microbiome and metabolome analysis.
  One vaginal swab for fetal fibronectin assessment will be taken at each study visit (total of three per participant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High risk singleton pregnancy for preterm birth
  Interventions: Device: Cervical stiffness assessment; Other: Cervical length measurement; Other: Fetal fibronectin

INTERVENTIONS:
Device: Cervical stiffness assessment — The cervical stiffness is assessed by using the licensed, CE-marked Pregnolia System, during a sterile speculum examination. The single-use, sterile Pregnolia Probe is placed on the anterior lip of the cervix at 12 o'clock position and a recording of cervical stiffness is generated over maximum 60 seconds (typically ̴15 seconds) and displayed as Cervical Stiffness Index (CSI) in mbar. The measurement is repeated 3 consecutive times without any time lag.
Other: Cervical length measurement — Cervical length measurement will be obtained via transvaginal ultrasound using a GE Voluson E10 ultrasound machine and 7.5MHz transvaginal probe. All measurements will be performed with the woman in a supine position with an empty bladder in the sagittal plane measuring from the internal to external cervical OS. The full length of the cervical canal will be visualized with the closed portion of cervix remaining being measured. Three measurements are taken with the shortest being documented as the final assessment.
Other: Fetal fibronectin — Vaginal swab collection. The specimen will be obtained from the posterior fornix over 10 seconds using the polyester tipped swab provided in the Hologic specimen collection kit. This sample will be then be stored frozen and processed using the Rapid fFN 10Q System (HOLOGIC, Marlborough, MA, USA) within 3 months.

SUMMARY:
Preterm birth (PTB), defined as delivery before 37 weeks gestation, is a common complication of pregnancy and affects up to 1 in 10 women in the UK. PTB is the leading cause of neonatal mortality and morbidity with babies born earliest being at the greatest risk. Identifying women at high risk of having a PTB and offering treatments and intervention to try and prevent this outcome is a huge priority in clinical practice and in government policy.

The PRECISION study will explore the use of a new antenatal test of cervical stiffness to try and improve the recognition of women who may deliver early. Current clinical practice involves measurement of cervical length (CL) and fetal fibronectin in women known to be high risk for PTB. However recent research suggests these methods could be improved upon and we may be able to recognise women at risk more reliably and at an earlier stage in the pregnancy if we use cervical stiffness assessments.

A licensed, CE-marked, vacuum-aspiration device called the Pregnolia system has been developed to give quantitative cervical stiffness index scores during pregnancy. This study will directly compare cervical length measurements and fetal fibronectin results with cervical stiffness, using the Pregnolia system, during the second trimester in women known to be high risk for preterm birth. The investigators will aim to explore the best possible predictive tool kit bundle for PTB using any combination of these assessments.

DETAILED DESCRIPTION:
PRECISION is a single site prospective, exploratory, cohort study of 60 women with a singleton pregnancy who are high risk for preterm birth.

Participants will have study assessments at 3 time points in second trimester as part of their routine care in high risk pre-term birth clinic. The study assessments will include transvaginal cervical length scanning, fetal fibronectin swabs and cervical stiffness assessment using the Pregnolia device.

Once recruited, participants will remain in the study until delivery and discharge from hospital. The investigators will collect routine clinical data from all participants' notes and electronic hospital records for maternal and neonatal outcomes. All study visits will coincide with routine care and all participating women will receive routine antenatal care throughout their pregnancy as per Saving Babies Lives Care Bundle V2, NICE Preterm Labour and Birth guideline and the North West Regional network preterm birth guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Singleton pregnancy
* Able to provide informed consent
* Meets criteria for high-risk pre-term birth clinic;

  * Previous PPROM <34+0 weeks
  * Previous sPTB <34+0 weeks
  * Previous spontaneous mid trimester miscarriage >16 weeks

Exclusion Criteria:

* Previous cervical surgery including previous trachelectomy, cone biopsy, loop excision or previous cerclage
* Existing cervical cerclage (vaginal or abdominal)
* Any cervical pathology at 12 o'clock position on cervix
* Vaginal bleeding evident on examination
* Visible, symptomatic cervical or vaginal infections
* Symptomatic of preterm birth (SROM, cervical dilatation)
* Known congenital uterine anomalies
* Known or suspected structural/chromosomal fetal abnormality
* Known HIV
* Cervical carcinoma
* Previous fully dilated emergency caesarean section
* Non-English speaking if unable to provide suitable verbal translation services (language line) at the time of recruitment or subsequent study visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female of reproductive age with confirmed singleton pregnancy.
Study Population: Participants will be recruited directly from the pre-term birth clinic at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with Spontaneous preterm birth <34 weeks gestation | Gestation at delivery.
  We will define sPTB as labour having occurred prior to 34+0 weeks of gestation in patients with either intact membranes or PPROM (<37 weeks). This excludes iatrogenic causes for preterm delivery including induction of labour (in the absence of PPROM) or elective caesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sharp, MBBS,BSc,PhD, Study Director — University of Liverpool
Locations (1):
- Liverpool Women's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medford E, Lane S, Sharp A, Care A. The PRECISION study protocol: Can cervical stiffness in the second trimester predict preterm birth in high-risk singleton pregnancies? A feasibility, cohort study. PLoS One. 2025 Feb 21;20(2):e0316297. doi: 10.1371/journal.pone.0316297. eCollection 2025. PMID 39982966
- See also: Cervical stiffness assessment device website — https://en.pregnolia.com/